CLINICAL TRIAL: NCT01432093
Title: Intensive Glycemic Management and Outcomes Following Liver Transplantation: A Randomized Controlled Trial
Brief Title: Intensive Glycemic Management and Outcomes Following Liver Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Gunjan Gandhi, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-002918
Record Dates: First submitted 2011-09-07; First posted 2011-09-12 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Hospital Hyperglycemia; Post-transplant Hyperglycemia
Keywords: liver transplant; high blood sugars; hospital hyperglycemia; post-transplant hyperglycemia; post liver transplant; post liver-kidney transplant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intensive glycemic management (Active Comparator): Multifaceted approach to achieve strict glucose goals of 90 to 120 mg/dL in the ICU and hospital wards.
  Interventions: Other: Intensive glycemic management
- Conventional management (Active Comparator): Conventional treatment to control hyperglycemia with a target glucose goal of 120 to 150 mg/dL in the ICU and 140 to 180 mg/dL on the hospital floors.
  Interventions: Other: Conventional management

INTERVENTIONS:
Other: Intensive glycemic management — Intravenous insulin infusion, strict dietary intervention, carbohydrate matched subcutaneous insulin therapy. This is a multifaceted approach to achieve strict glucose goals of 90 to 120 mg/dL in the ICU and hospital wards.
  Arms: Intensive glycemic management
Other: Conventional management — Conventional treatment to control hyperglycemia with a target glucose goal of 120 to 150 mg/dL in the ICU and 140 to 180 mg/dL on the hospital floors.
  Arms: Conventional management

SUMMARY:
Most people develop high blood sugars following liver transplant that requires treatment with insulin in the hospital, even if they don't have diabetes, due to stress and use of steroid medications. High blood sugar levels can be treated with a hormone that the body makes called insulin. This study is being done to determine if maintaining normal blood sugar levels after transplant for as long as needed while in the hospital results in a lesser incidence of death, infections, transplanted liver rejection or failure or need for rehospitalization within 90 days after transplant.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Undergoing liver transplant or combined liver-kidney transplant

Exclusion Criteria:

* Unable to grant informed consent or comply with study procedure
* Allergic to any of the excipients in insulin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2011-10; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Conduct a randomized controlled trial to compare outcomes with two management strategies to control hospital hyperglycemia in adult patients following liver transplantation. | 90 days following liver transplantation.
  The primary outcome is a 90 day composite of mortality by any cause, graft failure, rejection, infections, and rehospitalization following liver transplantation.

SECONDARY OUTCOMES:
Compare length of stay in the ICU and hospital in the two study groups. | 90 days following liver transplantation.
Compare the incidence of hypoglycemia in the ICU and hospital in the two study groups. | 90 days following liver transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Gunjan Y. Gandhi, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Jacksonville, Florida, United States